CLINICAL TRIAL: NCT04509596
Title: A Phase I, Open-Label, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of DZD1516 in Combination With Trastuzumab and Capecitabine, or DZD1516 in Combination With T-DM1, in Patients With Metastatic HER2 Positive (HER2+) Breast Cancer
Brief Title: DZD1516 in Combination With Trastuzumab and Capecitabine, or in Combination With T-DM1, in Patients With Metastatic HER2 Positive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2019HE001
Record Dates: First submitted 2020-08-03; First posted 2020-08-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer Metastatic
MeSH Terms: interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- daily dose of DZD1516 (Experimental): daily dose of DZD1516
  Interventions: Drug: DZD1516 mono therapy in Part A, DZD1516 in combination with trastuzumab and/or capecitabine in Part B, DZD1516 in combination with T-DM1 in Part C

INTERVENTIONS:
Drug: DZD1516 mono therapy in Part A, DZD1516 in combination with trastuzumab and/or capecitabine in Part B, DZD1516 in combination with T-DM1 in Part C — Part A is twice daily (except Cycle 0) oral dosing of DZD1516, starting from 50 mg. If tolerated, dose will be escalated in subsequent cohorts until MTD.
  Part B is twice daily oral dosing of DZD1516 in combination with capecitabine 1000 mg/m2 orally twice daily on Days 1-14 of each 21-day cycle or with trastuzumab 8 mg/kg intravenously (IV) on Day 1 of Cycle 1, followed by 6 mg/kg on Day 1 of each 21-day cycle.
  Part C is twice daily oral dosing of DZD1516 in combination with T-DM1 3.6 mg/kg intravenously (IV) once every 21 days

SUMMARY:
DZD1516 is an oral, blood brain barrier penetrable, selective HER2 tyrosine kinase inhibitor. This study is designed to evaluate the safety and tolerability of DZD1516 in patients with metastatic HER2 positive breast cancer who have progressed following prior therapy. This is the first time this drug has ever been tested in patients, and so it will help to understand what type of side effects may occur with the drug treatment. It will also measure the levels of drug in the body and assess its anti-cancer activity as monotherapy and in combination with trastuzumab and/or capecitabine, or in combination with T-DM1

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Male or female patients aged ≥ 18 years
* histologically or cytologically confirmed HER2 positive advanced breast cancer which failed prior therapies
* Predicted life expectancy ≥ 12 weeks.
* ECOG performance status 0 to 1 for patients without LM, and 0 to 2 for patients with LM at the time of signing ICF
* Adequate bone marrow reserve and organ system functions
* For patients without CNS metastases, patients must have at least one measurable lesion according to RECIST (version 1.1)
* For patients with Brain metastasis: Patient must have at least one measurable intracranial lesion according to modified RECIST 1.1

Exclusion Criteria:

* Intervention with any of the following: Any investigational agents or study drugs from a previous clinical study within 4 weeks of the first dose of study treatment； Any cytotoxic chemotherapy or other anticancer drugs for the treatment of metastatic breast cancer from a previous treatment regimen within 4 weeks of the first dose of study treatment； Any intrathecal chemotherapy within 2 weeks of the first dose of study treatment；Major surgery procedure (excluding placement of vascular access), or significant traumatic injury within 4 weeks of the first dose of study treatment, or have an anticipated need for major surgery during the study； Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment;
* CNS complications that require urgent neurosurgical intervention
* Any evidence of severe or uncontrolled systemic diseases
* Another malignancy within 5 years prior to enrolment with the exception of adequately treated in-situ carcinoma of the cervix, uterus, basal or squamous cell carcinoma or non-melanomatous skin cancer.
* Live vaccines within 4 weeks prior to first dose.
* Active infections including:Tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice)；Positive Hepatitis B surface antigen (HBsAg) or positive HCV antibodies or confirmed positive HIV test result.
* Refractory nausea and vomiting if not controlled by supportive therapy, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of DZD1516
* Involvement in the planning and conduct of the study (applies to Sponsor staff or staff at the study site).
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | up to approximately 1 year
  To investigate the safety and tolerability of DZD1516
Incidence of dose limiting toxicities (DLTs) | 21 days after the first multiple dose
  To investigate the safety and tolerability of DZD1516
To define maximum tolerated dose (MTD) of DZD1516 if possible (Part A only) | 21 days after the first multiple dose
  To investigate the safety and tolerability of DZD1516
To define Recommended Phase II Combination Dose (RP2CD) of DZD1516 in combination with trastuzumab and capecitabine (Part B only) | 21 days after the first multiple dose
  To investigate the safety and tolerability of DZD1516 in combination with either trastuzumab, capecitabine, or both trastuzumab and capecitabine
To define Recommended Phase II Combination Dose (RP2CD) of DZD1516 in combination with T-DM1 (Part C only) | 21 days after the first multiple dose
  To investigate the safety and tolerability of DZD1516 in combination with T-DM1

SECONDARY OUTCOMES:
Drug concentrations of DZD1516 and its metabolite DZ2678 in plasma, urine and CSF | up to approximately 6 months
  Pharmacokinetics endpoints
Maximum plasma concentration (Cmax) of DZD1516 and its metabolite DZ2678 | up to approximately 6 months
  Pharmacokinetics endpoints
Area under the plasma concentration-time curve (AUC) of DZD1516 and its metabolite DZ2678 | up to approximately 6 months
  Pharmacokinetics endpoints
Plasma concentration of capecitabine and metabolites 5-FU (Part B only) | up to approximately 6 months
  Pharmacokinetics endpoints
Plasma Cmax of capecitabine and 5-FU (Part B only) | up to approximately 6 months
  Pharmacokinetics endpoints
Plasma AUC of capecitabine and 5-FU (Part B only) | up to approximately 6 months
  Pharmacokinetics endpoints
Plasma concentration of DM1 (Part C only) | up to approximately 6 months
  Pharmacokinetics endpoints
Objective Response Rate (ORR) | up to approximately 1 year
  To assess preliminary anti-tumor efficacy of DZD1516 as monotherapy and as combination therapy
Disease Control Rate (DCR) | up to approximately 1 year
  To assess preliminary anti-tumor efficacy of DZD1516 as monotherapy and as combination therapy
Duration of Response (DoR) | up to approximately 1 year
  To assess preliminary anti-tumor efficacy of DZD1516 as monotherapy and as combination therapy
Progression free survival (PFS) (Part B and Part C on) | up to approximately 1 year
  To assess preliminary anti-tumor efficacy of DZD1516 as combination therapy
Overall survival (for patients with leptomeningeal metastasis in Part B and Part C only) | up to approximately 1 year
  To assess preliminary anti-tumor efficacy of DZD1516 as combination therapy

CONTACTS AND LOCATIONS:
Overall Officials: McAndrew, Principal Investigator — UCLA Hematology/Oncology Parkside
Locations (3):
- UCLA Hematology/Oncology Parkside, Santa Monica, California, United States
- China (2):
  - Zhejiang Cancer Hospital, Hangzhou
  - Cancer Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, McAndrew NP, Wang X, Du Y, DiCarlo B, Wang M, Chen K, Yu W, Hu X. Preclinical and clinical activity of DZD1516, a full blood-brain barrier-penetrant, highly selective HER2 inhibitor. Breast Cancer Res. 2023 Jul 6;25(1):81. doi: 10.1186/s13058-023-01679-4. PMID 37415239